CLINICAL TRIAL: NCT00315354
Title: Popular Diets, Metabolism, and CVD Risk
Brief Title: Popular Diets Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Professor, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DK072428 (NIH); R01DK072428 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Obesity; Insulin Resistance
Keywords: obesity; nutrition
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Diet, Fat-Restricted

ARMS (3):
- 1 (Experimental): Low glycemic index diet
  Interventions: Other: Low glycemic index diet
- 2 (Active Comparator): Low fat diet
  Interventions: Other: Low fat diet
- 3 (Active Comparator): Very low carbohydrate diet
  Interventions: Other: Very low carbohydrate diet

INTERVENTIONS:
Other: Low glycemic index diet — Feeding protocol, all foods prepared in a metabolic kitchen
  Arms: 1
Other: Low fat diet — Feeding protocol, all foods prepared in a metabolic kitchen
  Arms: 2
Other: Very low carbohydrate diet — Feeding protocol, all foods prepared in a metabolic kitchen
  Arms: 3

SUMMARY:
The aim of this study is to evaluate the effects of three dominant dietary patterns - conventional low-fat, low-glycemic index (GI) and very-low-carbohydrate - on energy metabolism and heart disease risk factors following weight loss in obese young adults in a feeding study

DETAILED DESCRIPTION:
For most of the last half century, reduction in fat intake has been the primary nutritional approach for the prevention and treatment of obesity and cardiovascular disease (CVD). Over the last few years, very low carbohydrate (Atkins-type) diets have achieved great popularity, with publication of several studies suggesting greater weight loss and improvements in CVD risk factors over 3 to 6 months. Recently, a third dietary approach focused on glycemic index (GI) has generated interest. However, few studies have compared the effects of these diets on body weight regulation and risk for CVD. The primary hypotheses of this study are that any diet that lowers the postprandial rise in blood glucose (very-low-carbohydrate or low-GI) will have beneficial effects on the physiological adaptations to weight loss and on some CVD risk factors. However, other CVD risk factors will be adversely affected by a very-low-carbohydrate vs. a low-GI diet. Preliminary data provide strong support for these hypotheses, by showing that resting energy expenditure declines less and CVD risk factors improve more with weight loss on a low-glycemic load diet compared to a conventional low-fat diet. This application proposes a cross-over feeding design to study the effects of three diets following 12.5% weight loss in obese young adult subjects (n = 24, age 18 to 40 years). The diets are: 1) conventional low-fat, with 60% carb, 20% fat, 20% protein; 2) low-GI with 40% carb, 40% fat, 20% protein; and 3) very-low-carbohydrate with 10% carb, 60% fat, 30% protein. The primary outcome is resting energy expenditure (indirect calorimetry). Secondary outcomes include total energy expenditure (doubly labeled water), thermic effect of food (indirect calorimetry), physical activity (accelerometry), insulin resistance and B-cell function (frequently-sampled OGTT), blood lipids, blood pressure and measures of systemic inflammation and coagulopathy. This study should have major public health implications to the millions of Americans currently following diets to decrease body weight and risk for heart disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2
* Willing and able to come to the GCRC 5 days per week to consume a supervised meal and pick-up food for all other meals
* Available for scheduled hospital admissions
* Willing to abstain from alcohol consumption for the duration of the study
* If female, regular menstrual cycles (defined as 26 to 30 days between cycles; no more than one day variation in the duration of menstrual flow)

Exclusion Criteria:

* Weight > 350 lbs
* Change in body weight (± 10%) over preceding year
* Taking any medications or dietary supplements that might affect body weight, appetite, or energy expenditure
* Smoking (1 cigarette in the last week)
* High levels of physical activity
* Currently following a special diet
* Abnormal laboratory screening tests
* Type 2 diabetes mellitus
* Allergies or aversions to foods on the study menu
* Previous diagnosis of an eating disorder or any other mental health disorder
* If female, pregnant in the past 12 months or planning to become pregnant during the study period
* If female, lactating in the preceding 12 months
* If taking birth control medication, change in medication in previous 3 months or plans to change medication during the study period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
resting energy expenditure using indirect calorimetry in the fasting state | end of each dietary period
insulin resistance assessed by frequently-sampled oral glucose tolerance test | end of each dietary period
thyroid function tests | end of each dietary period

SECONDARY OUTCOMES:
total energy expenditure using doubly labeled water methodology | end of each dietary period
thermic effect of food using indirect calorimetry | end of each dietary period
physical activity using accelerometry | end of each dietary period
serum lipids | end of each dietary period
plasminogen activator inhibitor-1 | end of each dietary period
C-reactive protein | end of each dietary period
blood pressure | end of each dietary period
hunger/appetite | end of each dietary period
insulin 30 minutes after oral glucose (as an effect modifier) | baseline
Core temperature | End of each dietary period
secreted frizzle-related protein-4 | end of each dietary period
heme-oxygenase | end of each dietary period
Irisin | end of each dietary period
fibroblast growth factor-21 | end of each dietary period
chemerin | end of each dietary period
trimethylamine N-oxide | fasting and postprandial, end of each dietary period
alanine aminotransferase | end of each dietary period
Uric acid | end of each dietary period
insulin | fasting and postprandial, end of each dietary period
ghrelin | fasting and postprandial, end of each dietary period
gastric inhibitory peptide | fasting and postprandial, end of each dietary period
GLP1 | fasting and postprandial, end of each dietary period
PYY | fasting and postprandial, end of each dietary period
Amylin | fasting and postprandial, end of each dietary period
Leptin | end of each dietary period
Metabolomic analysis | end of each dietary period
  Evaluate the effect of diet on metabolomic profile in plasma, with the aim of assessing dietary adherence and exploring diet-disease mechanisms

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Cara B Ebbeling, PhD, Study Director — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Walsh CO, Ebbeling CB, Swain JF, Markowitz RL, Feldman HA, Ludwig DS. Effects of diet composition on postprandial energy availability during weight loss maintenance. PLoS One. 2013;8(3):e58172. doi: 10.1371/journal.pone.0058172. Epub 2013 Mar 6. PMID 23483989
- [Result] Ebbeling CB, Swain JF, Feldman HA, Wong WW, Hachey DL, Garcia-Lago E, Ludwig DS. Effects of dietary composition on energy expenditure during weight-loss maintenance. JAMA. 2012 Jun 27;307(24):2627-34. doi: 10.1001/jama.2012.6607. PMID 22735432
- [Derived] Angelidi AM, Bartell E, Huang Y, Zeleznik OA, Estanyol-Torres N, Mi MY, Bhupathiraju SN, Kelly RS, Wittenbecher C, Lasky-Su J, Clish CB, Ludwig DS, Ebbeling CB, Hirschhorn JN. Weight-independent effects of dietary carbohydrate-to-fat ratio on metabolomic profiles: secondary outcomes of a 5-month randomized controlled feeding trial. Nat Commun. 2026 Jan 17. doi: 10.1038/s41467-026-68353-z. Online ahead of print. PMID 41547934
- [Derived] Hron BM, Ebbeling CB, Feldman HA, Ludwig DS. Hepatic, adipocyte, enteric and pancreatic hormones: response to dietary macronutrient composition and relationship with metabolism. Nutr Metab (Lond). 2017 Jul 5;14:44. doi: 10.1186/s12986-017-0198-y. eCollection 2017. PMID 28694840
- [Derived] Esko T, Hirschhorn JN, Feldman HA, Hsu YH, Deik AA, Clish CB, Ebbeling CB, Ludwig DS. Metabolomic profiles as reliable biomarkers of dietary composition. Am J Clin Nutr. 2017 Mar;105(3):547-554. doi: 10.3945/ajcn.116.144428. Epub 2017 Jan 11. PMID 28077380